CLINICAL TRIAL: NCT02561013
Title: A Randomized, Controlled, Clinical Study to Assess a New Adjustable Compression Device in Patients With Venous Leg Ulcers
Brief Title: A Clinical Study to Assess a Compression Device in Patients With Venous Leg Ulcers
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business reasons
Sponsor: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-013293
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Varicose Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3M™ Coban™ Custom Fit Compression System (Experimental): 3M™ Coban™ Custom Fit Compression System will be custom-fitted at first subject visit and will thereafter be applied and removed daily by the study subject. It will be worn throughout the day by the study subject and removed before bedtime. It will provide therapeutic compression for edema control to help in the healing of venous leg ulcers.
  Interventions: Device: 3M™ Coban™ Custom Fit Compression System
- Profore (Active Comparator): Profore multi-layer compression bandaging system will be applied at the first subject visit and will be worn by the study subject continuously for 7 days, at which time it will be replaced with a new system, or, in the case of a product or non-product reason, replaced before 7 days. It will provide therapeutic compression for edema control to help in the healing of venous leg ulcers
  Interventions: Device: Profore

INTERVENTIONS:
Device: 3M™ Coban™ Custom Fit Compression System — 3M Coban™ Fit is a compression system that consists of two components: 1. A Compression Stocking and 2. Coban™ Fit Sleeve.
  The stocking provides compression to the foot and improves wearing comfort in the calf area under the sleeve. The compression sleeve is intended to provide the therapeutic compression to the calf, with the initial fitting to be done by a health-care professional. The compression sleeve is customized according to the anatomy of the patient's leg; both components are designed to be used together.
  Other Names: Coban Fit Compression System
  Arms: 3M™ Coban™ Custom Fit Compression System
Device: Profore — PROFORE is a multi-layer compression bandaging system developed to apply sustained graduated compression for the management of venous leg ulcers and associated conditions. Multi-layer compression bandaging is the first choice in treatment for venous leg ulcers.
  Arms: Profore

SUMMARY:
The purpose of this study is to evaluate the product performance of a new adjustable compression system for the treatment of venous leg ulcers.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the product performance of a new adjustable compression system for the treatment of venous leg ulcers. The new compression system consists of a compression stocking and and adjustable compression sleeve. It will be used over primary dressings to provide compression that is beneficial to the healing of venous leg ulcers.

ELIGIBILITY:
Inclusion Criteria:

1. Is the subject 21 years or older?
2. Does the subject have an active venous leg ulceration? If multiple ulcers are present, the investigator will need to select a single ulcer of the study leg that is > 2cm apart from any other ulcer?
3. Does the subject have an ulcer size between 1cm2 and 12cm2?
4. Does the subject have an ABPI between 0.8 and 1.3 that was taken within the past 28 days?
5. Is the subject ambulatory?
6. Is the subject or family member willing to self-manage the venous leg ulcer therapy at home in collaboration with the medical staff, including the ability to properly readjust the closure straps as indicated by tension indicators, and apply new dressings when needed?
7. Is the subject able to understand questionnaire items and action items (e.g., Subject Diary)?
8. Is the subject willing to give written informed consent, including permission to take photographs of the study leg?

Exclusion Criteria:

1. Does the subject have severe arterial occlusive disease?
2. Does the subject have decompensated heart insufficiency NYHA Class IV, ACC.AHA Stage D?
3. Does the subject have septic phlebitis?
4. Does the subject have severe deep vein thrombosis (phlegmasia cerulea dolens) and other conditions contraindicated according to established guidelines and local procedures?
5. Does the subject have known hypersensitivity to any of the component materials?
6. Does the subject have a suspected clinical infection of the ulcer or any other systemic infection (requiring antibiotics)?
7. Is the subject scheduled for surgery for the ulcer during the 12 weeks following inclusion?
8. Does the subject have a hospital stay planned for the 12 weeks following inclusion?
9. Does the subject have a suspected or confirmed cancerous ulceration?
10. Does the subject have severe peripheral sensitive neuropathy?
11. Is the subject participating in any other prospective study interfering with this study?
12. Does the subject have any medical condition which in the professional opinion of the investigator disqualifies the subject from enrollment into the study?
13. Does the subject have a history of noncompliance to therapies?

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the number of ulcers achieving complete closure (100% epithelialization) after 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Wound area reduction and relative wound area reduction at weeks 4, 8, and 12. | Up to 12 weeks
Relative wound area reduction >/= 40% at Week 4 | 4 weeks
Time to complete closure | 1-12 weeks
Occurrence of treatment-related adverse events | 0-12 weeks
Occurrence of treatment-related drop-outs | 0-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J Parks, MD, PhD, Study Director — 3M Critical & Chronic Care Division
Locations (5):
- United States (3):
  - Institute for Advanced Wound Care, Montgomery, Alabama
  - HealthEast Care System, Saint Paul, Minnesota
  - Jobst Vascular Institute, Toledo, Ohio
- Canada (2):
  - Lawson Health Research Institute, London, Ontario
  - Calea Ltd, Mississauga, Ontario